CLINICAL TRIAL: NCT05108428
Title: MRI Guided Adaptive Radiation for Locally Advanced Rectal Adenocarcinoma to Enhance Complete Response
Brief Title: Adaptive Radiation for Locally Advanced Rectal Adenocarcinoma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Viewray Inc. (Industry); Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20911
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Rectal Adenocarcinoma
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms | interventions — Capecitabine; Radiotherapy; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRI-guided adaptive radiation (Experimental): Patients will receive capecitabine-based chemoradiotherapy (chemotherapy with capecitabine + radiation). Dosing will be modified based on tumor changes measured daily and weekly by MR-guided radiotherapy (MRgRT) utilizing MR-linac (MRL) systems. Chemoradiotherapy will be followed by standard of care consolidated chemotherapy. (FOLFOX)
  Interventions: Drug: Capecitabine; Radiation: Radiation Therapy; Drug: FOLFOX regimen

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 825 mg/m^2 twice daily orally 5 days per week on days of planned radiation therapy.
  Other Names: Xeloda
Radiation: Radiation Therapy — Participants will receive varying doses of radiotherapy based on MRI guidance, beginning at 28-33 fractions (1.8 Gray units) .
Drug: FOLFOX regimen — Standard of Care FOLFOX regimen consists of 8 cycles (each cycle is 14 days) of 5-fluorouracil, leucovorin, and oxaliplatin. Dosage is as follows: Oxaliplatin 85 mg/m^2 IV over 2 hours day 1 each cycle. Leucovorin (optional) 400 mg/m^2 IV over 2 hours day 1 each cycle. 5-fluorouracil bolus* (optional) 400 mg/m^2 IV push day 1 of each cycle, and 5-fluorouracil infusion 2400 mg/m^2 IV continuous infusion over 46 hours day 1 each cycle.

SUMMARY:
The purpose of the study is to determine the feasibility of using magnetic resonance imaging (MRI)-guided adaptive chemoradiation therapy to improve response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance status of 0, 1
* Histologically confirmed diagnosis of adenocarcinoma of the rectum.
* Clinical Stage II or III as determined on rectal MRI with a distal tumor extent/margin no more than 1 cm proximal to the anterior peritoneal reflection.
* Must have the ability to swallow and retain oral medications
* Adequate hematologic function within 28 days before registration as defined in protocol.
* Adequate hepatic function within 45 days before registration, as defined in protocol.
* Adequate renal function within 28 days before registration, as defined in protocol.
* International normalized ratio of prothrombin time (INR) and prothrombin time (PT) within 28 days before registration must be within normal limits for the lab. Patients who are therapeutically treated with an agent such as warfarin may participate if they are on a stable dose and no underlying abnormality in coagulation parameters exists per medical history
* Pregnancy test done within 14 days before registration must be negative (for women of childbearing potential only). Pregnancy testing should be performed according to institutional standards.

Exclusion Criteria:

* Patients with one or more of the following conditions are NOT eligible for this study:
* Rectal cancer histology other than adenocarcinoma (i.e., sarcoma, lymphoma, squamous cell carcinoma, mucosal melanoma, mixed adenoneuroendocrine, anal adenocarcinoma, etc.).
* History of prior invasive rectal malignancy, regardless of disease-free interval or history of familial polyposis syndrome (Lynch, FAP, etc.).
* Patients with a history of antineoplastic treatment for prior malignancy within the past 3 years, except for adequately treated basal cell skin carcinoma or in situ cervical cancer. Note: Hormone therapy for breast cancer is permitted.
* Primary unresectable rectal cancer. Note: A tumor is considered unresectable when invading adjacent organs and an en bloc resection will not achieve negative margins.
* Synchronous colorectal adenocarcinomas.
* Tumor may not be causing symptomatic bowel obstruction
* Definitive clinical or radiologic evidence of metastatic disease or nodal disease outside of the prescribed radiation field. Note: Required imaging studies must have been performed within 28 days prior to enrollment.
* Patients with a history of an arterial thrombotic event within the past 6 months. This includes angina (stable or unstable), myocardial infarction, transient ischemic attack (TIA), Cardiovascular Accident (CVA). Note: Patients with a history of venous thrombotic episodes such as deep venous thrombosis, pulmonary embolus occurring more than 6 months prior to enrollment may be considered for protocol participation, provided they are on stable doses of anticoagulant therapy. Similarly, patients who are anticoagulated for atrial fibrillation or other conditions may participate, provided they are on stable doses of anticoagulant therapy.
* No other experimental therapies (including chemotherapy, radiation, hormonal treatment, antibody therapy, immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, matric metalloprotease inhibitors, thalidomide, anti-VEGF (vascular endothelial growth factor) monoclonal antibody or other experimental drugs) of any kind are permitted while the patient is receiving study treatment.
* Inflammatory bowel disease or have a history of abdominal surgery that may interfere with gastrointestinal motility or absorption.
* Ineligibility to undergo MR imaging or treatment on the MRL due to medical or physical reasons. Anxiety disorders will be permitted if pre-medicated with anxiolytics.
* Active seizure disorder uncontrolled by medication.
* Major surgery within 12 weeks before enrollment.
* Any prior pelvic radiation.
* Known DPD (dihydro pyrimidine dehydrogenase) deficiency. Any of the following because this study involves agents that have known or potential genotoxic or mutagenic and teratogenic effects: Pregnant women, Nursing women who are unwilling to discontinue nursing, Men or women of childbearing potential who are unwilling to employ adequate contraception (e.g. hormonal or barrier method of birth control; abstinence) for the duration of study treatment and for 3 months after the last dose of study therapy.
* Any diagnosis of acquired immunodeficiency syndrome (AIDS-related illnesses) or known human immunodeficiency virus (HIV) disease.
* Co-morbid illnesses or other concurrent disease that, in the judgement of the clinician obtaining informed consent, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens or prevent required follow-up.
* BMI > 40 is considered exclusive from this study due to increased surgical complication risk and greater risk of incomplete resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of MRI guided dose adaptive chemoradiation therapy | Up to 6 weeks
  Investigators will demonstrate if MRI guided dose-adaptation based on MR morphologic objective measurements during primary chemoradiation is feasible. Feasibility will be recorded for each patient as an indicator variable (1=feasible; 0=not feasible)

SECONDARY OUTCOMES:
Number of Participants with Complete Clinical Response (cCR) | Up to 6 months
  Complete Clinical Response is defined as the absence of clinically detectable tumor after treatment.
Number of Participants with Pathological Complete Response (pCR) | Up to 6 months
  Pathological Complete Response (pCR) is defined as the lack of all signs of cancer in tissue samples after treatment.

OTHER OUTCOMES:
Number of Participants with Disease-Free Survival (DFS) | Up to 5 years
  Disease-free survival is defined as the length of time after primary treatment ends that the patient survives without any signs or symptoms of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Frakes, MD, Principal Investigator — Moffitt Cancer Center; Seth Felder, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No